CLINICAL TRIAL: NCT06517342
Title: E-lombaqual: Motivations, Obstacles and Opportunities for Using a Health Application to Encourage Physical Activity in People With Chronic Low Back Pain
Brief Title: Motivations, Obstacles and Opportunities for Using a Health Application to Encourage Physical Activity in People With Chronic Low Back Pain
Acronym: E-lombaqual
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2024 LECHAUVE
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low-back Pain
Keywords: chronic low back pain; m-health; smartphone; qualitative study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In industrialized countries, low back pain can be considered a priority health issue. Some studies define it as one of the leading causes of disability in people under 45, or the leading cause of musculoskeletal disorders, with a prevalence of 26.9%. Chronic forms account for less than 10% of acute episodes, but represent around 85% of costs. It has been recognized that rest and physical inactivity are not beneficial in the treatment of low back pain, and worse, increase the risk of chronicity. Functional Restoration of the Spine (FRS) programs have been introduced in rehabilitation centers, and have proved to be effective both physically and psycho-socially. Patients generally adhere well to this type of program during in-center treatment. The effects obtained tend to fade rapidly on discharge, due to a lack of adherence to what can be offered conventionally (exercise sheets, oral advice). The development of connected tools (smartphones, tablets, etc.) could be a lever in this respect, as it would enable better patient support. In 2022, 84% of the population will own a smartphone. The content offered would be of higher quality, and would enable regular remote monitoring of the patient. The effects of the initial intensive treatment would be maintained by this new interactive, fun tool.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Chronic non-specific low-back pain.
* Diagnosis confirmed according to HAS definition (i.e. pain located between the thoraco-lumbar hinge and the lower gluteal fold. It may be associated with radiculalgia corresponding to pain in one or both lower limbs at the level of one or more dermatomes). Patients included in the study must have given written informed consent.

Exclusion Criteria:

* Patients not meeting HAS diagnostic criteria
* Patients with comprehension difficulties (making it impossible to fill in questionnaires)
* Patients with medical contraindications to physical exercise
* Patients under guardianship, curatorship or safeguard of justice.
* Patients without a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be contacted in the Physical Medicine and Rehabilitation department of Clermont-Ferrand University Hospital for a presentation of the study. They will be given an information leaflet and time to reflect on their participation. If the patient agrees to take part, the EAPA will schedule an appointment to complete the non-objection form. A semi-structured interview will be scheduled in an office on the PRM ward, in order to meet the study objectives. Again, the objectives of the study will be stated, as well as the instructions for this structured interview.
  Questionnaires will be submitted and completed only after the interview. Data will be collected on a dictaphone and then manually transcribed into text format (verbatims) during the interview by a second operator.
  An a posteriori analysis will be carried out using the qualitative method. The interview guide is likely to be adapted according to the first individual interviews, as required by the qualitative method.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Phenomenological analysis of semi-structured interviews with patients. | Up to 1 day
  45-minute semi-structured interview

SECONDARY OUTCOMES:
Identification of patient expectations via a semi-structured interview | Up to 1 day
  45-minute semi-structured interview
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : sex in ration Male and femalle
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : age in year
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : height in cm
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : family situation as a couple or single
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : weight in Kg
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : level of education (no diploma, less than baccalaureate, baccalaureate or more than baccalaureate)
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : lifestyle (active, retired, disabled)
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : living environment (urban, rural)
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : regular physical activity (frequency, type of activity)
Characterization of patients' profiles using a socio-demographic | Up to 1 day
  Responses to the socio-demographic questionnaire : leisure activities (frequency, type)
Physical Activity Perception Scale | Up to 1 day
  Self-questionnaire score: Physical Activity Perception Scale (EPAP). Identification of barriers and levers to regular physical activity using the EPAP questionnaire. This questionnaire contains 26 items on the facilities and obstacles encountered when engaging in physical activity. The maximum score for this questionnaire is 100 points thanks to an equation. Responses range from "Strongly disagree" (0 points) to "Strongly agree" (4 points). The total score ranges from 0 - "Poor perception of physical activity" to 100 - "Excellent perception of physical activity".
Visual Analogue Pain Scale | Up to 1 day
  Visual Analogue Pain Scale (VAS Pain). A value of 10 indicates very intense pain. On the contrary, a pain value of 0 means that no pain is felt.
Functional disability | Up to 1 day
  Self-questionnaire score: OSWESTRY Disabitity Index (ODI). Questionnaire on disability rated by a Likert scale ranging from 0 "no restriction" to 5 "severe restriction". scores can range from 0 to 50 points. a score of 0 to 4 indicates no disability. A score of 5 to 14 indicates a mild disability, 15 to 24 a moderate disability, and 25 to 34 a severe disability. A higher score indicates complete disability.
Fears and beliefs | Up to 1 day
  Self-questionnaire score : Fear Avoidance Belief Questionnaire (FABQ). The FABQ consists of 2 subscales, corresponding to two distinct subsections. The first subscale (items 1-5) is the physical activity subscale (FABQPA; PA - Physical activity), and the second subscale (items 6-16) is the work subscale (FABQW; W-Work). Each subscale is ranked separately by summing the item responses of the respective scale (0-6 for each item). For scoring purposes, only 4 of the physical items on the activity scale are rated (24 possible points) and only 7 of the work items (42 possible points). A higher score indicates higher levels of fear-avoidance beliefs.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No